CLINICAL TRIAL: NCT05709327
Title: Integrating Smart Ring Wearable Technology in Pregnancy Health Monitoring (I-SMART)
Acronym: I-SMART
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Principal Investigator, Tan Kok Hian, Professor, KK Women's and Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2021/2515
Record Dates: First submitted 2022-12-26; First posted 2023-02-02 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Pregnancy

STUDY DESIGN:
Intervention Model Description: Single-arm observational study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single-arm observational study (Other): All participants in the study will be provided a smart ring to wear for the entire duration of the pregnancy.
  Interventions: Other: Integrating Smart Ring Wearable Technology in Pregnancy Health Monitoring (I-SMART)

INTERVENTIONS:
Other: Integrating Smart Ring Wearable Technology in Pregnancy Health Monitoring (I-SMART) — Single-arm observational study where all participants in the study will be given a smart ring (Oura Ring) to wear throughout the duration of the study.

SUMMARY:
This study aims to test the following hypotheses in a single-arm observational study in 70-100 healthy pregnant multi-ethnic women who will be followed-up from the first trimester of pregnancy to the third trimester of pregnancy.

Aim 1: To assess the applicability, acceptability and compliance with the use of a wearable smart ring together with smart digital devices (e.g., smart phone) during pregnancy.

Hypothesis 1: The investigators hypothesize that participants will respond favorably to the use of the smart ring to monitor their physical activity and sleep during pregnancy.

Aim 2: To assess the association between maternal characteristics (age, pre-pregnancy BMI, pregnancy weight gain, stress, anxiety and depression symptoms) with physical activity markers (energy expenditure, and step count) and sleep markers (duration, quality, sleep onset latency, wake after sleep onset, time in bed and heart rate variability) collected from the smart ring in the second trimester of pregnancy.

Hypothesis 2: The investigators hypothesize that specific maternal characteristics will be associated with physical activity markers (energy expenditure, and step count), as well as sleep markers (duration, quality, sleep onset latency, wake after sleep onset, time in bed and heart rate variability).

DETAILED DESCRIPTION:
Wearable sensor and other smart technologies may play an important part in the early detection of adverse pregnancy-related health events along with motivating improvement in patient and provider interactions for effective pregnancy health management. The use of wearable sensors, more specifically, wearable smart rings can potentially be used to offer remote, unobtrusive personalized care, encourage preventive care and provide the necessary context for self-help based just-intime adaptive interventions (feedback loops utilizing digital phenotyping data to trigger in-app interventions). Studies on the use of wearable smart rings and health outcomes are scarce, and currently there is no available data of the use of wearable smart rings together with smart digital devices (i.e., smart phone) for tracking pregnancy health in women. This study aims to be the first to generate preliminary pilot data to support it's use in this specific group of women.

An observational period for up to 37 weeks, single-center, one-armed intervention study involving 70-100 healthy pregnant women from a multi-ethnic population (Chinese, Malay, Indian, others) aged between 21 and 45 years.

All participants included into the study will be provided an Oura Ring to wear for the rest of the pregnancy period.

Data will be collected through questionnaires and each time a participant opens up their mobile application, the uploaded data will be automatically transferred via Bluetooth connection to the study database in the smart ring cloud service. The questionnaires include socio-economic factors, maternal anxiety and depression, maternal sleep, and maternal physical activity. The participants data will be collected from the moment join the study up till delivery.

ELIGIBILITY:
Inclusion criteria:

1. From the first to third trimester of pregnancy (4-39 weeks of gestational age)
2. Mobile phone's operating system supported by the smart ring application.
3. Aged 21 and above

Exclusion criteria:

1. Can't read or speak English
2. Below 21 years of age
3. Below or above gestational age limit
4. Limited mobility
5. Diagnosed with severe unstable mental conditions
6. Diagnosed with severe chronic disorders
7. Mobile device not compatible with smart ring

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy pregnant women
Enrollment: 100 (Estimated)
Dates: Start 2023-09-03 (Actual); Primary Completion 2025-12-03 (Estimated); Study Completion 2025-12-03 (Estimated)

PRIMARY OUTCOMES:
Feasibility and applicability of smart ring usage during pregnancy | At the end of pregnancy
  The feasibility and applicability of a commercial smart ring (Oura Ring) use assessed by a feedback survey.

SECONDARY OUTCOMES:
Objective change in sleep quality across the entire pregnancy | up to 37 weeks from recruitment
  The smart ring (Oura Ring) will issued to capture durations of deep sleep, rapid eye movement (REM) sleep, light sleep and nightly heart rate. Sleep Score ranges from 0-100, where a higher score reflects better sleep outcome.
Self-reported change in sleep quality | First trimester of pregnancy between 0-12 weeks gestational age
  Self-reported sleep quality will be assessed using the Pittsburgh Sleep Quality Index. Total score ranging from 0 to 21 with the higher total score (referred to as global score) indicating worse sleep quality.
Self-reported change in sleep quality | Second trimester of pregnancy between 13-27 weeks gestational age
  Self-reported sleep quality will be assessed using the Pittsburgh Sleep Quality Index. Total score ranging from 0 to 21 with the higher total score (referred to as global score) indicating worse sleep quality.
Self-reported change in sleep quality | Third trimester of pregnancy between 28-40 weeks gestational age
  Self-reported sleep quality will be assessed using the Pittsburgh Sleep Quality Index Questionnaire (PSQI). Total score ranging from 0 to 21 with the higher total score (referred to as global score) indicating worse sleep quality.
Objective change in physical activity across the entire pregnancy | up to 37 weeks from recruitment
  The smart ring (Oura Ring) will be issued to capture durations of activity, inactivity and rest. Activity score ranges from 0-100, where a higher score reflects better balance between activity and rest.
Self-reported change in physical activity | First trimester of pregnancy between 0-12 weeks gestational age
  Self-reported physical activity will be assessed using the International Physical Activity Questionnaire (IPAQ). Data collected with International Physical Activity Questionnaire (IPAQ) can be reported as a continuous measure and reported as median metabolic equivalent of task (MET) minutes. A higher score will indicated higher physical activity involvement.
Self-reported change in physical activity | Second trimester of pregnancy between 13-27 weeks gestational age
  Self-reported physical activity will be assessed using the International Physical Activity Questionnaire (IPAQ). Data collected with International Physical Activity Questionnaire (IPAQ) can be reported as a continuous measure and reported as median metabolic equivalent of task (MET) minutes. A higher score will indicated higher physical activity involvement.
Self-reported change in physical activity | Third trimester of pregnancy between 28-40 weeks gestational age
  Self-reported physical activity will be assessed using the International Physical Activity Questionnaire (IPAQ). Data collected with International Physical Activity Questionnaire (IPAQ) can be reported as a continuous measure and reported as median metabolic equivalent of task (MET) minutes. A higher score will indicated higher physical activity involvement.
Anxiety and depression symptoms | First trimester of pregnancy between 0-12 weeks gestational age
  The Depression Anxiety Stress Scales (DASS) will be used to capture self-reported anxiety and depression symptoms across pregnancy. The minimum score is 0 and the maximum score is 63. A higher score on the DASS indicates greater severity or frequency of these negative emotional symptoms.
Change in anxiety and depression symptoms across the first, second and third trimesters | Second trimester of pregnancy between 13-27 weeks gestational age
  The Depression Anxiety Stress Scales (DASS) will be used to capture self-reported anxiety and depression symptoms across pregnancy. The minimum score is 0 and the maximum score is 63. A higher score on the DASS indicates greater severity or frequency of these negative emotional symptoms.
Change in anxiety and depression symptoms across the first, second and third trimesters | Third trimester of pregnancy between 28-40 weeks gestational age
  The Depression Anxiety Stress Scales (DASS) will be used to capture self-reported anxiety and depression symptoms across pregnancy. The minimum score is 0 and the maximum score is 63. A higher score on the DASS indicates greater severity or frequency of these negative emotional symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Kok Hian Tan, MD, Principal Investigator — KK Women's and Children's Hospital
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-12-19): https://cdn.clinicaltrials.gov/large-docs/27/NCT05709327/Prot_SAP_000.pdf